CLINICAL TRIAL: NCT02897999
Title: A Placebo-Controlled, Blinded, Dose-Escalation, Study to Assess the Safety and Pharmacodynamics of Single and Multiple Doses of QBKPN (Inactivated Klebsiella Pneumoniae) Site Specific Immunomodulator (SSI), Administered Subcutaneously to Healthy Male and Female Volunteers
Brief Title: Single and Multiple Dose Evaluation of QBKPN SSI In Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Qu Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QBKPN-03
Record Dates: First submitted 2016-08-19; First posted 2016-09-13 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- SAD Cohort 1 (Experimental): Single dose of 0.05 mL QBKPN or Placebo
  Interventions: Biological: QBKPN; Other: Placebo
- SAD Cohort 2 (Experimental): Single dose of 0.10 mL QBKPN or Placebo
  Interventions: Biological: QBKPN; Other: Placebo
- SAD Cohort 3 (Experimental): Single dose of 0.20 mL QBKPN or Placebo
  Interventions: Biological: QBKPN; Other: Placebo
- SAD Cohort 4 (Experimental): Single dose of 0.40 mL QBKPN or Placebo
  Interventions: Biological: QBKPN; Other: Placebo
- SAD Cohort 5 (Experimental): Single dose of 0.80 mL QBKPN or Placebo
  Interventions: Biological: QBKPN; Other: Placebo
- SAD Cohort 6 (Experimental): Single dose of 1.2 mL QBKPN or Placebo
  Interventions: Biological: QBKPN; Other: Placebo
- MAD Cohort 1 (Experimental): 5 doses of QBKPN or Placebo administered every other day (using one of the dose from the SAD Cohort)
  Interventions: Biological: QBKPN; Other: Placebo
- MAD Cohort 2 (Experimental): 5 doses of QBKPN or Placebo administered every other day (using one of the dose from the SAD Cohort)
  Interventions: Biological: QBKPN; Other: Placebo
- MAD Cohort 3 (Experimental): 5 doses of QBKPN or Placebo administered every day (using one of the dose from the SAD Cohort)
  Interventions: Biological: QBKPN; Other: Placebo
- MAD Cohort 4 (Experimental): 5 doses of QBKPN or Placebo administered every day (using one of the dose from the SAD Cohort)
  Interventions: Biological: QBKPN; Other: Placebo

INTERVENTIONS:
Biological: QBKPN — QBKPN Site Specific Immunomodulators
Other: Placebo — Placebo

SUMMARY:
The purpose of this dose-escalation study is to assess the safety and pharmacodynamics of single and multiple doses of QBKPN SSI, administered subcutaneously to healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking (at least for 6 months prior to first study drug administration) males or females, 18 to 65 years of age, inclusive at the time of informed consent.
* Body mass index (BMI) that is within 18.5 - 30.0 kg/m2, inclusive.
* Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination
* Systolic blood pressure between 95-140 mmHg, inclusive, and diastolic blood pressure between 55-90 mmHg, inclusive, and heart rate between 50-100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
* QTc interval ≤ 450 milliseconds for males and females, unless deemed otherwise Not Clinically Significant by the Principal Investigator/Sub-Investigator.
* Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
* Agree not to have a tattoo or body piercing until the end of the study.
* Agree to practice effective methods of contraception

Exclusion Criteria:

* Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.
* A known history or positive test result for human immunodeficiency virus (HIV), chronic Hepatitis B surface antigen, or Hepatitis C.
* A positive test result for drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), alcohol test and cotinine. Positive pregnancy test for female subjects.
* Known history or presence of (1) Alcohol abuse or dependence within one year prior to first study drug administration; (2) Drug abuse or dependence; (3) Known or suspected hypersensitivity to any component of the product (4) Food allergies and/or presence of any dietary restrictions; or (5) Severe allergic reactions (e.g. anaphylactic reactions, angioedema).
* Recent history (within 8 weeks prior to screening) of travel to or emigration from any country with high incidence for tuberculosis.
* A positive tuberculin skin (PPD) test result

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse events [Safety and Tolerability] | 2 weeks
  Incidence, severity, and dose-relationship of adverse events, vital signs, and clinical laboratory parameters

SECONDARY OUTCOMES:
Changes in cellular biomarkers over time | 2 weeks
  Absolute (#/mL) and Differentials (%)
Immunological biomarkers analysis | 2 weeks

OTHER OUTCOMES:
MAD Cohorts only: Changes in cell surface markers on neutrophils and monocytes over time | 2 weeks
MAD cohorts only: Gene Expression Analysis | 2 weeks
Phenotype and Genotype Correlation [Exploratory gene association analysis] | 2 weeks